CLINICAL TRIAL: NCT02874586
Title: Plasma Exchange Combination of Immunosuppressive Regimens for the Remission of Auto-immune Hepatitis
Brief Title: Plasma Exchange Combination of Immunosuppressive Regimens for Auto-immune Hepatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaoli Fan (Other)
Responsible Party: Sponsor-Investigator, Xiaoli Fan, Principal Investigator, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIH-2
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Hepatitis, Autoimmune
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Plasma exchange combination of immunosuppressive regimens (Experimental): Plasma exchange(once) ,with the following standard immunosuppressive regimens for the remission of auto-immune hepatitis
  Interventions: Other: Plasma exchange combination of immunosuppressive regimens

INTERVENTIONS:
Other: Plasma exchange combination of immunosuppressive regimens

SUMMARY:
An open-label,pilot study to evaluate the efficacy and safety of plasma exchange combination of immunosuppressive regimens, for the remission of autoimmune hepatitis (AIH).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with auto-immune hepatitis based on liver biopsy results, with the indications of immunosuppressive therapy;
* High levels of total bilirubin (TB) (≥10 X ULN);
* High levels of immunoglobulin G(IgG) (≥1.5 X ULN);
* Agreed to participate in the trial, and assigned informed consent;

Exclusion Criteria:

* The presence of hepatitis A, B, C, D, or E virus infection;

  * Patients with presence of liver cirrhosis or portal hypertension;
  * Primary sclerosing cholangitis, non-alcoholic steatohepatitis, drug induced liver disease or Wilson disease confirmed by liver biopsy;
  * Pregnant and breeding women;
  * Patients with severe anemia (hemoglobin < 8 g/dL), leukopenia (WBC < 2500/mm3), or thrombocytopenia (platelet count < 50,000/mm3);
  * Severe disorders of other vital organs, such as severe heart failure, cancer;
  * Parenteral administration of blood or blood products within 6 months before screening;
  * Recent treatment with drugs having known liver toxicity;
  * Taken part in other clinic trials within 6 months before screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2021-04 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Percent of patients that achieve biochemical remission of AIH | Month 6 after the treatment initiated

SECONDARY OUTCOMES:
Alanine transaminase (ALT) | Day 1, and Week 1, 2, 4, 12, 24
Aspartate transaminase(AST) | Day 1, and Week 1, 2, 4, 12, 24
Globin(GLB) | Day 1, and Week 1, 2, 4, 12, 24
Immunoglobulin G(IgG) | Day 1, and Week 1, 2, 4, 12, 24
Total bilirubin(TB) | Day 1, and Week 1, 2, 4, 12, 24
Direct bilirubin(DB) | Day 1, and Week 1, 2, 4, 12, 24

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, MD, Study Chair — West China Hospital,Chengdu, Sichuan, China
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided